CLINICAL TRIAL: NCT01800903
Title: Clinical Study Investigating Safety and Performance of a New Coating for Urinary Intermittent Catheters in Healthy Volunteers
Brief Title: Safety and Performance of a New Coating for Urinary Intermittent Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CP235; CP235 (Other: Coloplast)
Record Dates: First submitted 2013-02-22; First posted 2013-02-28 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Intermittent Urethral Catheterization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sequence 1 (Active Comparator): SpeediCath catheter then ZN-D catheter then ZN-C catheter
  Interventions: Device: ZN-D catheter; Device: ZN-C catheter; Device: SpeediCath catheter
- Sequence 2 (Experimental): SpeediCath catheter then ZN-C catheter then ZN-D catheter
  Interventions: Device: ZN-D catheter; Device: ZN-C catheter; Device: SpeediCath catheter
- Sequence 3 (Experimental): ZN-D catheter then SpeediCath catheter then ZN-C catheter
  Interventions: Device: ZN-D catheter; Device: ZN-C catheter; Device: SpeediCath catheter
- Sequence 4 (Experimental): ZN-D catheter then ZN-C catheter then SpeediCath catheter
  Interventions: Device: ZN-D catheter; Device: ZN-C catheter; Device: SpeediCath catheter
- Sequence 5 (Experimental): ZN-C catheter then SpeediCath catheter then ZN-D catheter
  Interventions: Device: ZN-D catheter; Device: ZN-C catheter; Device: SpeediCath catheter
- Sequence 6 (Experimental): ZN-C catheter then ZN-D catheter then SpeediCath catheter
  Interventions: Device: ZN-D catheter; Device: ZN-C catheter; Device: SpeediCath catheter

INTERVENTIONS:
Device: ZN-D catheter — ZN-D catheter is a catheter, similar to the CE-marked SpeediCath, but with a newly developed coating.
Device: ZN-C catheter — ZN-C catheter is a catheter, similar to the CE-marked SpeediCath, but with a newly developed coating.
Device: SpeediCath catheter — The Speedicath cathere is CE-marked and commercially available.

SUMMARY:
The aim of the study is to evaluate safety and performance of a new catheter coating,compared to the current SpeediCath coating.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and signed letter of authority
2. Be at least 18 years of age and have full legal capacity
3. Be a male
4. Willing to refrain from using analgetics up to 24 hours prior to catheterization visits

Exclusion Criteria:

1. Abnormalities, diseases or surgical procedures performed in the lower urinary tract
2. Symptoms of urinary tract infections (at least one of the following: frequent urination, stinging or pain at urination)
3. Participating in other interventional clinical investigations during this investigation (inclusion to termination) or have previously participated in this investigation (including run-in period)
4. Known hypersensitivity toward any of the test products -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, MD, PhD, Principal Investigator — Department of Urology, Rigshospitalet Denmark
Locations (1):
- Department of Urology, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 subjects were included in the safety population. 4 subjects discontinued because they were unable to catheterize with given catheter. these drop-outs were distributed evenly among the catheter types:
  1. subject: ZN-C
  2. subjects: ZN-D
  1 subjects: SC
  These subjects were excluded from the ITT population as no endpoints were registered for them
Groups:
- SpeediCath Catheter Then ZN-D Catheter Then ZN-C Catheter: First SpeediCath catheter then ZN-D catheter then ZN-C catheter
- SpeediCath Catheter Then ZN-C Catheter Then ZN-D Catheter: First SpeediCath catheter then ZN-C catheter then ZN-D catheter
- ZN-D Catheter Then SpeediCath Catheter Then ZN-C Catheter: First ZN-D catheter then SpeediCath catheter then ZN-C catheter
- ZN-D Catheter Then ZN-C Catheter Then SpeediCath Catheter: First ZN-D catheter then ZN-C catheter then SpeediCath catheter
- ZN-C Catheter Then SpeediCath Catheter Then ZN-D Catheter: First ZN-C catheter then SpeediCath catheter then ZN-D catheter
- ZN-C Catheter Then ZN-D Catheter Then SpeediCath Catheter: First ZN-C catheter then ZN-D catheter then SpeediCath catheter
Period: First Test Period
Arm/Group | SpeediCath Catheter Then ZN-D Catheter Then ZN-C Catheter | SpeediCath Catheter Then ZN-C Catheter Then ZN-D Catheter | ZN-D Catheter Then SpeediCath Catheter Then ZN-C Catheter | ZN-D Catheter Then ZN-C Catheter Then SpeediCath Catheter | ZN-C Catheter Then SpeediCath Catheter Then ZN-D Catheter | ZN-C Catheter Then ZN-D Catheter Then SpeediCath Catheter
Started | 7 | 6 | 4 | 7 | 6 | 6
Completed | 7 | 6 | 4 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Test Period
Arm/Group | SpeediCath Catheter Then ZN-D Catheter Then ZN-C Catheter | SpeediCath Catheter Then ZN-C Catheter Then ZN-D Catheter | ZN-D Catheter Then SpeediCath Catheter Then ZN-C Catheter | ZN-D Catheter Then ZN-C Catheter Then SpeediCath Catheter | ZN-C Catheter Then SpeediCath Catheter Then ZN-D Catheter | ZN-C Catheter Then ZN-D Catheter Then SpeediCath Catheter
Started | 7 | 6 | 4 | 7 | 6 | 6
Completed | 6 | 6 | 4 | 7 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — unable to catheterise | 1 | 0 | 0 | 0 | 0 | 0
Period: Third Test Period
Arm/Group | SpeediCath Catheter Then ZN-D Catheter Then ZN-C Catheter | SpeediCath Catheter Then ZN-C Catheter Then ZN-D Catheter | ZN-D Catheter Then SpeediCath Catheter Then ZN-C Catheter | ZN-D Catheter Then ZN-C Catheter Then SpeediCath Catheter | ZN-C Catheter Then SpeediCath Catheter Then ZN-D Catheter | ZN-C Catheter Then ZN-D Catheter Then SpeediCath Catheter
Started | 6 | 6 | 4 | 7 | 6 | 6
Completed | 6 | 6 | 4 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: The intention to treat population consists of 36 healthy male subjects
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Discomfort During Catheterization
Description: Evaluated by the subject on a 10 cm Visual Analog Scale (VAS), where 0 cm is no discomfort and 10 cm is the worst possible discomfort.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: cm
Groups:
- ZN-D Catheter: Subjects who tested the ZN-D catheter
- ZN-C Catheter: Subjects who tested the ZN-C catheter
- SpeediCath: Subjects who tested the Speedicath catheter
Arm/Group | ZN-D Catheter | ZN-C Catheter | SpeediCath
Number analyzed (Participants) | 35 | 35 | 36
cm | 2.6 (2.2) | 2.4 (1.7) | 1.8 (1.5)

ADVERSE EVENTS:
Groups:
- All Participants: Data from subjects in the safety population. Definition of safety population: subjects that have given informed consent and have been exposed to at least one product.
  However for 4 of these subjects no endpoint data was obtained and they were not included in the ITT population; they therefore do not appear in the participant flow module.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No